CLINICAL TRIAL: NCT05378347
Title: Endurant Stent Graft System vs Excluder Endoprothesis: A Global, Prospective, Randomized Clinical Trial in Sac Regression
Brief Title: Endurant Stent Graft System vs Excluder Endoprothesis: ADVANCE Trial
Acronym: ADVANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDT21033
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Abdominal Aortic Aneurysm; Abdominal Aortic Aneurysm >= 5.5 Centimeters in Male (Disorder); Abdominal Aortic Aneurysm >= 5.0 Centimeters in Female (Disorder)
Keywords: EVAR, AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical Events Committee members as well as key sponsor team members will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Medtronic Endurant II/IIs (Experimental): Subjects are randomized on a 1:1 basis to receive an EVAR procedure with either a Medtronic Endurant II/IIs endoprothesis or Gore's Excluder / Excluder Conformable.
  Interventions: Device: Medtronic Endurant II or Endurant IIs Stent Graft System
- Gore Excluder / Excluder Conformable (Experimental): Subjects are randomized on a 1:1 basis to receive an EVAR procedure with either a Medtronic Endurant II/IIs endoprothesis or Gore's Excluder / Excluder Conformable.
  Interventions: Device: Gore Excluder or Gore/ Excluder Conformable AAA Endoprosthesis

INTERVENTIONS:
Device: Medtronic Endurant II or Endurant IIs Stent Graft System — EVAR treatment with Medtronic Endurant II/IIs Stent Graft System
  Arms: Medtronic Endurant II/IIs
Device: Gore Excluder or Gore/ Excluder Conformable AAA Endoprosthesis — EVAR treatment with Excluder / Excluder Conformable Stent Graft System
  Arms: Gore Excluder / Excluder Conformable

SUMMARY:
The purpose of this trial is to generate clinical evidence related to key performance outcomes of Endurant II/IIs Stent Graft Systems verses Gore Excluder / Excluder Conformable AAA Endoprosthesis in subjects with Abdominal Aortic Aneurysms. Subjects are randomized and imaging collected at all follow-up time points to assess the primary endpoint.

DETAILED DESCRIPTION:
This is a post-market, prospective, interventional, global, multi-center, randomized, dual-arm clinical trial. The primary objective of this trial is to evaluate sac regression outcomes of the Medtronic Endurant II/IIs Stent Graft System and Gore Excluder/Excluder Conformable AAA Endoprosthesis in standard EVAR subjects. Subjects are randomized on a 1:1 basis to receive EVAR with either a Medtronic Endurant II/IIs Stent Graft Systems or Gore Excluder / Excluder Conformable AAA Endoprosthesis. Data is collected pre- and post-procedure at discharge, at 30 days, and once a year until the 5-year follow-up is completed. An estimate of 550 subjects (minimum 500) are enrolled at up to 100 sites globally, with the potential to extend enrollment up to 900 subjects based on predictive probability analysis to adequately achieve either non-inferiority or superiority for the primary endpoint.

Product Names:

* Medtronic Endurant II/IIs Stent Graft System
* Gore Excluder and/or Gore Excluder Conformable AAA Endoprosthesis Imaging is collected for all follow-up time points and are evaluated by a core lab for the key primary and secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Subject and the treating physician agree that the subject will return for all required followup visits
* Subject or legal representative or consultee, as applicable, has consented for trial participation and signed the Informed Consent approved by the sponsor and by the Ethics Committee/Institutional Review Board
* Subject has an aneurysm diameter of ≥ 5 cm (if woman) ≥ 5.5 cm (if man)
* Subject's AAA anatomy is appropriate for both Medtronic Endurant II/IIs Stent Graft System and Gore Excluder/Excluder Conformable AAA Endoprosthesis as per assessment of both treating physician and Core Lab in accordance with the overlapping commercially available IFUs per applicable region.

Exclusion Criteria:

* Subject is participating in an investigational drug or device study which may bias or interfere with the endpoints and follow-up of this trial
* Subject has an estimated life expectancy of ≤ 3 years as judged by the investigator
* Subject has an aneurysm that is:

  1. Suprarenal/pararenal/juxtarenal
  2. Isolated ilio-femoral
  3. Mycotic
  4. Inflammatory
  5. Pseudoaneurysm
  6. Concomitant or prior dissection involving the abdominal aorta or iliac arteries
  7. Ruptured
  8. Symptomatic AAA
* Subject has significant thrombus and / or calcium at the arterial implantation sites, specifically the proximal aortic neck and distal iliac artery interface. Significant thrombus may be quantified as thrombus ≥ 2 mm in thickness and / or ≥ 25% of the vessel circumference in the intended seal zone of the aortic neck.
* Subject requires emergent aneurysm treatment, for example, trauma or rupture
* Subject with connective tissue disease that may have caused the aneurysm e.g. Marfan syndrome, Ehlers-Danlos, Loeys-Dietz syndrome
* Subject has previously undergone surgical or endovascular treatment in the abdominal aorta or the iliac arteries for aneurysm or occlusive disease
* Planned use of aorto-uni-iliac (AUI) main body device
* Any planned additional device (apart from the main body, limb stent graft and extensions per assigned treatment per randomization) during index or staged procedure, e.g., endostaple or anchor, Iliac branch endoprosthesis, embolization, etc.
* Planned coverage of the internal iliac artery/arteries
* Subject has an estimated glomerular filtration rate (eGFR) < 45 ml/min/1.73m2 or subject is on dialysis
* Subject has a systemic infection who may be at increased risk of endovascular graft infection, per investigator's discretion
* Subject has a psychiatric or other condition that may interfere with the trial, per investigator's discretion
* Subject is of childbearing potential in whom pregnancy cannot be excluded
* Subject has a known hypersensitivity or contraindication to anticoagulants, anti-platelets, or contrast media, which is not amenable to pre-treatment
* Subject belongs to a vulnerable population per investigator's judgment
* Subject has an active COVID-19 infection or relevant history of COVID- 19

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subject has an aneurysm diameter of ≥ 5 cm (if woman) ≥ 5.5 cm (if man)
Enrollment: 550 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Sac Regression | 12 months
  Proportion of patients with sac regression at 1 year, defined in accordance with SVS guidelines as the reduction in maximum diameter by >= 5 mm when compared to the first CT imaging study obtained within 90 days after index procedure.

SECONDARY OUTCOMES:
Aneurysm sac change by diameter as a continuous variable | 12 months and annually to 5 years
Aneurysm sac change by volume incidence rate | 12 months and annually to 5 years
Type II endoleak incidence rate | 30 days, 12 months and annually to 5 years
Type I endoleak incidence rate | 30 days,12 months and annually to 5 years
Secondary intervention incidence rate | 30 days, 12 months and annually to 5 years
All cause mortality incidence rate | 30 days, 12 months and annually to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schermerhorn, MD, Principal Investigator — Beth Israel Deaconess Medical Center, United States; Hence Verhagen, MD, Principal Investigator — Erasmus University Medical Center, Netherlands
Locations (67):
- United States (32):
  - Loma Linda University Medical Center, Loma Linda, California
  - Hoag Hospital, Newport Beach, California
  - University of California Irvine Medical Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Francisco UCSF Medical Center, San Francisco, California
  - Denver Health Medical Center, Denver, Colorado
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Northside Hospital Forsyth, Atlanta, Georgia
  - Northshore University Health System, Skokie, Illinois
  - Ascension Via Christi Saint Francis, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - VA Maryland Health Care System, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Albany Medical College, Albany, New York
  - Northwell Health Lenox Hill Hospital, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - University Hospitals, Cleveland Medical Center, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Cardiovascular Surgery Clinic, Memphis, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
- France (4):
  - Assistance Publique - Hopitaux de Marseille Hopital de la Timone, Marseille, Marseille Cedex
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hospices Civils de Lyon-CHU Lyon, Lyon
  - Hopital de Hautepierre - CHU de Strasbourg, Strasbourg
- Germany (7):
  - University Hospital Augsburg, Augsburg
  - University Hospital Cologne, Cologne
  - Elisabeth Hospital Essen, Essen
  - Universitatsklinikum Frankfurt, Frankfurt
  - University Hospital Leipzig, Leipzig
  - University Hospital rechts der Isar of the Technical University Munich, Munich
  - St. Franziskus Hospital Munster, Münster
- University Hospital of Larisa, Larissa, Greece
- Italy (3):
  - Fondazione IRCCS Ca' Granda - Ospendale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - AOU Citta della Salute e della Scienza di Torino, Torino
- Japan (5):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Niigata University Medical and Dental Hospital, Chuo Ku, Niigata
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Keio University Hospital, Shinjuku-Ku, Tokyo
- Netherlands (4):
  - Rijnstate Hospital, Arnhem, The Netherlands
  - Amsterdam University Medical Center, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Erasmus Medisch Centrum, Rotterdam
- Hospital Universitario Son Espases, Palma, Mallorca, Spain
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Luzerner Kantonsspital, Lucerne
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (2):
  - Oxford University Hospitals NHS Trust - John Radcliffe Hospital, Oxford, Oxfordshire
  - Royal Infirmary of Edinburgh, Edinburgh